CLINICAL TRIAL: NCT02950740
Title: Evaluation of Nutritional Status, Food Intake and Fecal Microbiota of 1-3 Year-old Children From Four Regions of Brazil
Brief Title: Nutritional Status, Food Intake and Fecal Microbiota of Brazilians Toddlers
Acronym: Nutrilife
Status: Completed | Type: Observational
Sponsor: Danone Early Life Nutrition Brazil (Industry)
Collaborators: Faculdade de Medicina do ABC (Other); Universidade Federal do Rio Grande do Norte (Other); Universidade Federal do Triangulo Mineiro (Other); Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Karina Vieira de Barros Munhoz, Health Care Nutrition Science Manager, Danone Early Life Nutrition Brazil
Other Study IDs: DanoneELN-01
Record Dates: First submitted 2016-03-31; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Child Nutrition Disorders
Keywords: malnutrition
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood sample (plasma, serum and erythrocytes Fecal sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Center 01 (SA): Toddlers from Santo André Early Childhood Public School
- Center 02 (POA): Toddlers from Porto Alegre Early Childhood Public School
- Center 03 (MG): Toddlers from Uberaba Early Childhood Public School
- Center 04 (RN): Toddlers from Natal Early Childhood Public School

SUMMARY:
Food intake pattern and lifestyle are associated with the nutritional status and intestinal microbiota composition, and such factors are important for the proper growth and development during early childhood, as well as for the health throughout life. This cross-sectional and multicenter study will include a total of 200 children aged between 1-3 years, enrolled in early childhood public schools from different regions of Brazil (Santo André, Uberaba, Porto Alegre and Natal). Data on birth and gestational history will be collected in a form. Nutritional status will be assessed by determining the weight and height, with subsequent calculations and classification of nutritional indices. A single blood sample will be collected to investigate the blood levels of vitamins A and D, iron, calcium, alkaline phosphatase and zinc, and feces will be collected for intestinal microbiota analysis. Food intake will be assessed by direct weighing of food in 2 non-consecutive days. Considering the importance of a well-balanced diet and its effects on the child's growth, development and intestinal colonization, this study purpose is to investigate potential associations among food intake, nutritional status and intestinal microbiota of early childhood infants from four regions of Brazil.

DETAILED DESCRIPTION:
It is a cross-sectional and multicenter study to examine two hundred children aged between 1-3 years, duly enrolled under full-time regimen in public schools of the cities of Santo André (SP), Uberaba (MG), Porto Alegre (RS) and Natal (RN). The Principal Site of study will be Fundação de Medicina do ABC, located in the city of Santo André, while Universidade Federal do Triângulo Mineiro, Universidade Federal of Ciências da Saúde de Porto Alegre and Universidade Federal do Rio Grande do Norte will be the other Sites. For such purpose, fifty children from each Early Childhood Public School will be screened according to the inclusion criteria and invited to participate in the study. Each State may include more than one Institution, if required to reach the total number of children established previously.

After the authorization and signature of the Informed Consent Form - ICF - (Attachment I) are given by the mother or legal responsible, such person must go to the Institution on the scheduled date for the collection of a blood sample and to deliver of a stool sample, collected as per prior orientation. The interviewer shall complete a questionnaire to obtain information on the birth and gestational history and current information on the child. A single blood sample will be collected for analysis of vitamins A and D, calcium, iron, ferritin, hemoglobin, zinc, selenium, alkaline phosphatase and lipids (cholesterol - total and fractions - and triglycerides), and a stool sample will be collected for analysis of parasites and microbiota in the feces.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 1-3 years
* Enrolled under full-time regimen in public schools
* Without any acute infection at the time of data collection.

Exclusion Criteria:

* Any chronic disease or congenital malformation
* Use of antibiotics in the past 30 days.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 200 children aged between 1-3 years, under full-time regimen in public schools of four cities of Brazil (Santo André, Uberaba, Porto Alegre and Natal). Fifty children of each city will be evaluated.
Sampling Method: Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Child Nutritional disorders | up to two months
  Obesity, overweight

SECONDARY OUTCOMES:
Levels of blood cells | up to three months
  laboratory parameters: blood count
Fatty acids composition | up to three months
  analysis in erythrocytes
Microbiota | up to three months
  Diversity of fecal microbiota
deficiency of minerals | up to three months
  laboratory parameters: calcium, zinc, selenium
Deficiency of retinol | up to three months
  Laboratory parameters: blood retinol
Levels of alkaline phosphatase | up to three months
  Laboratory parameters:alkaline phosphatase
Levels of ferritin | up to three months
  Laboratory parameters: ferritin
Deficiency of vitamin D | up to three months
  Laboratory parameters:level of vitamin D
Food intake | up to two months
  Direct food weighing
Problems in child growth | up to two months
  stunting

IPD SHARING:
Plan to Share IPD: No